CLINICAL TRIAL: NCT00750854
Title: A Double Arm Study to Evaluate the Effectiveness of NEM Compositions for the Treatment of Joint and Connective Tissue Pain
Brief Title: Efficacy & Safety Study of Natural Eggshell Membrane (NEM) for the Treatment of Joint & Connective Tissue Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ESM Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CLN# C0104
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis; Fibromyalgia
Keywords: arthritis; osteoarthritis; fibromyalgia; connective tissue disorder
MeSH Terms: conditions — Osteoarthritis; Fibromyalgia; Arthritis; Connective Tissue Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEM Treatment 1 (Experimental): NEM Formulation X (#0802), 500 mg, once daily, orally
  Interventions: Dietary Supplement: NEM Formulation X
- NEM Treatment 2 (Experimental): NEM Formulation Y (#0505), 500 mg, once daily, orally
  Interventions: Dietary Supplement: NEM Formulation Y

INTERVENTIONS:
Dietary Supplement: NEM Formulation X — see Treatment Arms
  Other Names: Natural Eggshell Membrane
  Arms: NEM Treatment 1
Dietary Supplement: NEM Formulation Y — see Treatment Arms
  Other Names: Natural Eggshell Membrane
  Arms: NEM Treatment 2

SUMMARY:
The purpose of this study was to evaluate the use of the dietary supplement Natural Eggshell Membrane (NEM) for the treatment of joint and connective tissue discomfort & pain.

DETAILED DESCRIPTION:
It is estimated that 140 million adults in the U.S. suffer from some form of joint or connective tissue (JCT) disorder (i.e. arthritis, lupus, gout, fibromyalgia, neck or back pain, etc.). As the population ages, this estimate is expected to grow rapidly. Traditional treatments for most of these disorders attempt to address only the symptoms (pain, inflammation, and discomfort) associated with the diseases. This usually involves the use of analgesics (i.e. acetaminophen, oxycodone, propoxyphene) or non-steroidal anti-inflammatory drugs (NSAIDs) (i.e. ibuprofen, diclofenac, celecoxib), alone or in combination. Most of these treatments have shown limited effectiveness in randomized controlled clinical trials (RCTs) or are known to have significant and sometimes severe side effects. To avoid the cardiac risks, gastrointestinal issues , and dependency issues associated with traditional JCT treatments (particularly with long-term use), many patients have turned to complementary and alternative medicines (CAMs) such as dietary supplements.

Glucosamine, chondroitin, and methylsulfonylmethane (MSM) alone and in combination, are widely marketed as dietary supplements to treat joint pain due to osteoarthritis (OA). Other vitamins, minerals, and botanicals such as kava, pine bark extract, capsicum, boswellia root extract, turmeric/curcumin, etc. are also marketed for various JCT pain maladies. We present here the use of eggshell membrane as a possible new natural therapeutic for JCT disorders. A single center, open label human clinical study was conducted to evaluate the efficacy and safety of NEM® as a treatment for pain associated with joint and connective tissue disorders. Subjects were to take NEM, 500mg, once daily for 30 days. Subjects were then evaluated for pain.

ELIGIBILITY:
Inclusion Criteria:

* patients seeking relief of mild to moderate pain due to joint or connective tissue (JCT)disorders.
* subjects must have had persistent pain associated with a JCT disorder.
* subjects were required to suspend all current pain relief medications.
* Subjects that were currently taking analgesic medications were eligible to participate in the studies following a 14 day washout period for NSAIDs, a 7 day washout for narcotics, and a 90 day washout for injected steroids.
* subjects currently taking glucosamine, chondroitin sulfate or MSM were only eligible after a 3-month washout period.

Exclusion Criteria:

* Patients were excluded if they were currently receiving remission-inducing drugs such as methotrexate or immunosuppressive medications or had received them within the past 3 months.
* body weight 250 pounds or greater.
* a known allergy to eggs or egg products.
* pregnant or breastfeeding women.
* subjects previously enrolled in a study to evaluate pain relief within the past 6 months or currently involved in any other research study involving an investigational product (drug, device, or biologic) or a new application of an approved product, within 30 days of screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-11; Primary Completion 2004-02 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure of this study was to evaluate the mean effectiveness of NEM® in relieving general pain associated with moderate Joint & Connective Tissue disorders. | 7 & 30 days

SECONDARY OUTCOMES:
A secondary objective of the study was to evaluate tolerability and any adverse reactions associated with supplementation with NEM®. | 7 & 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Leu, D.Ph., N.D., Principal Investigator; Kevin J Ruff, Ph.D., MBA, Study Director — ESM Technologies, LLC
Locations (1):
- Leu Private Practice, Jenks, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruff KJ, DeVore DP, Leu MD, Robinson MA. Eggshell membrane: a possible new natural therapeutic for joint and connective tissue disorders. Results from two open-label human clinical studies. Clin Interv Aging. 2009;4:235-40. doi: 10.2147/cia.s5797. Epub 2009 Jun 9. PMID 19554094
- See also: Study published in Clinical Interventions in Aging — http://www.dovepress.com/articles.php?article_id=3142